CLINICAL TRIAL: NCT06260124
Title: Acute Effects of Greek Traditional Dancing on Health, Performance and Muscle Damage Markers in Pre- and Postmenopausal Women: Implications of Dancing Tempo.
Brief Title: Acute Physiological Effects of Greek Traditional Dancing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Dimitrios Draganidis, Assisstant Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Greek Dancing-UTH
Record Dates: First submitted 2024-01-16; First posted 2024-02-15 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-01

CONDITIONS: Menopause; Cardiovascular Health; Body Composition; Physical Performance; Muscle Damage
Keywords: Greek traditional dancing; premenopausal women; postmenopausal women; dancing tempo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-menopausal women (Experimental): Pre-menopausal healthy, inactive women that will participate in a random order in three dancing sessions (Greek traditional dancing) of different tempo on non-consecutive days.
  Interventions: Other: Slow tempo; Other: Moderate tempo; Other: Fast tempo
- Post-menopausal (Experimental): Post-menopausal healthy, inactive women that will participate in a random order in three dancing sessions (Greek traditional dancing) of different tempo on non-consecutive days.
  Interventions: Other: Slow tempo; Other: Moderate tempo; Other: Fast tempo

INTERVENTIONS:
Other: Slow tempo — A single Greek traditional dance of slow tempo lasting 3-4 minutes.
Other: Moderate tempo — A single Greek traditional dance of moderate tempo lasting 3-4 minutes.
Other: Fast tempo — A single Greek traditional dance of fast tempo lasting 3-4 minutes.

SUMMARY:
In Greece, people of different age groups, including young children to older adults, are involved in traditional dance. To date, the well-know benefits of dancing include entertainment, socialization and increased physical activity. However, the acute effects of Greek traditional dancing on health, physical performance and muscle damage indices remain largely unknown. Therefore, the aim of this project is to evaluate the acute effect of Greek traditional dancing on health-, physical performance-, and muscle damage-related parameters by considering the impact of dancing tempo (slow vs moderate vs fast). In a crossover repeated measures design 10 pre- and 10 post-menopausal women will participate in the three dancing sessions of different tempo in a random order.

DETAILED DESCRIPTION:
This study aims at determining the acute effect of Greek traditional dancing on health- and physical performance-related parameters by considering the impact of dancing tempo. Ten pre- and ten postmenopausal women meeting the inclusion criteria will be assigned to a crossover trial. Initially, participants will undergo baseline testing including (i) anthropometrics, (ii) body composition, (iii) physical performance, (iv) physical activity level and (v) dietary intake. After baseline measurements, a 7-day familiarization period will take place, during which participants will practice daily on the three experimental dances. Each dance will be characterized by a different tempo (beats per minute) so that there will be one dance from each tempo category (i.e. slow, moderate and fast). After familiarization, participants will execute in a random order the three dancing sessions, on separate days. Each dancing session will consist of one dance (of either slow or moderate or fast tempo) lasting ~ 3- 4 minutes. During each dance heart rate, oxygen consumption and activity intensity will be continuously monitored. Before and immediately after the dance systolic and diastolic blood pressure, perceived exertion and blood lactate will be measure. In addition, before each dance and at 24 and 48 hours post-dance muscle soreness, muscle strength and resting metabolic rate will be measured and a resting blood sample will be drawn for the assessment of inflammatory and oxidative stress markers.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal and postmenopausal women.
* Abstain from vigorous physical activity and/or exercise during the last (at least) 6 months prior to the study.
* Free of musculoskeletal diseases and injuries.
* Free of cardiometabolic diseases.
* Free of mental health disorders
* No body weight loss >10% over the last 6 months prior to the study
* Non-smokers

Exclusion Criteria:

* Perimenopause and menopause women
* Participation vigorous physical activity and/or exercise during the last (at least) 6 months prior to the study
* Presence of musculoskeletal diseases and injuries.
* Presence of cardiometabolic diseases.
* Presence of mental health disorders
* Body weight loss >10% over the last 6 months prior to the study
* Smokers

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy pre-menopausal and post-menopausal women
Enrollment: 20 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | At baseline and immediately after the dance
  Systolic and diastolic blood pressure will be measured using a blood pressure cuff
Change in perceived exertion | At baseline and immediately after the dance
  Perceived exertion will be rated using the Borg Rating of Perceived Exertion scale, a numerical scale that ranges from 6 (no exertion) to 20 (maximum effort).
Change in blood lactate | At baseline and immediately after the dance
  Blood lactate will be measured on a portable, automatic lactate analyser using the relevant strips
Change in resting metabolic rate | At baseline and at 24 hours and 48 hours after the dance
  Resting metabolic rate (kcal) will be assessed using a portable open-circuit indirect calorimeter with a ventilated hood system
Change in delayed-onset of muscle soreness (DOMS) | At baseline and at 24 hours and 48 hours after the dance
  DOMS of the knee extensors and flexors of both limbs will be evaluated by palpation of the relaxed muscle's belly and distal region with participants rating the perceived soreness on a visual analogue scale ranging from 1 to 10.
Change in maximal isometric voluntary contraction | At baseline and at 24 hours and 48 hours after the dance
  Maximal isometric voluntary contraction of the knee extensors and flexors of both limbs will be assessed using an isokinetic dynamometer.
Change in joint range of motion | At baseline and at 24 hours and 48 hours after the dance
  Knee joint range of motion will be assessed using a manual goniometer
Change in functional performance | At baseline and at 24 hours and 48 hours after the dance
  Functional performance will be assessed using the movement-based screening tool functional movement screen (FMS)
Change in white blood cell count | At baseline and at 24 hours and 48 hours after the dance
  White blood cell count will be measured using an automatic blood analyzer
Change in granulocyte count | At baseline and at 24 hours and 48 hours after the dance
  Granulocyte count will be measured using an automatic blood analyzer
Change in lymphocytes | At baseline and at 24 hours and 48 hours after the dance
  Lymphocytes will be measured using an automatic blood analyzer
Change in monocytes | At baseline and at 24 hours and 48 hours after the dance
  Monocytes will be measured using an automatic blood analyzer
Change in creatine kinase concentration | At baseline and at 24 hours and 48 hours after the dance
  Creatine kinase will be measured using an automatic blood analyzer and commercially available kits
Change in reduced glutathione | At baseline and at 24 hours and 48 hours after the dance
  Reduced glutathione will be measured spectrophotometrically in red blood cells
Change in oxidized glutathione | At baseline and at 24 hours and 48 hours after the dance
  Oxidized glutathione will be measured spectrophotometrically in red blood cells
Change in catalase activity | At baseline and at 24 hours and 48 hours after the dance
  Catalase activity will be measured spectrophotometrically in red blood cells
Change in protein carbonyls | At baseline and at 24 hours and 48 hours after the dance
  Protein carbonyls will be measured spectrophotometrically in red blood cells
Change in total antioxidant capacity | At baseline and at 24 hours and 48 hours after the dance
  Total antioxidant capacity will be measured spectrophotometrically in plasma
Change in heart rate | Through dance session completion, an average of 30 minutes
  Heart rate will be continuously monitored using heart rate sensors
Change in oxygen consumption | Through dance session completion, an average of 30 minutes
  Oxygen consumption will be continuously monitored using a portable metabolic system.
Change in physical activity | Through dance session completion, an average of 30 minutes
  The number of steps performed will be assessed using an accelerometer (ActiGraph Gt3x)

SECONDARY OUTCOMES:
Change in red blood cell count | At baseline and at 24 hours and 48 hours after the dance
  Red blood cell count will be measured using an automatic blood analyzer
Change in hematocrit | At baseline and at 24 hours and 48 hours after the dance
  Hematocrit will be measured using an automatic blood analyzer
Change in hemoglobin | At baseline and at 24 hours and 48 hours after the dance
  Hemoglobin will be measured using an automatic blood analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Draganidis, PhD, Principal Investigator — University of Thessaly, Department of Physical Education and Sport Science
Locations (1):
- University of Thessaly, Department of Physical Education and Sport Science, Trikala, Thessaly, Greece